CLINICAL TRIAL: NCT03808376
Title: PROMISE Study: A Prospective, Multicenter Evaluation of Accuracy and Safety of an Implantable Continuous Glucose Sensor Lasting up to 180 Days
Brief Title: PROMISE Study: An Evaluation of an Implantable Continuous Glucose Sensor up to 180 Days
Acronym: PROMISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Senseonics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTP-0036
Record Dates: First submitted 2019-01-15; First posted 2019-01-17 (Actual); Results first posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-07

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Continuous Glucose Monitoring Device (Experimental): The Eversense® 180 CGM System
  Interventions: Device: Continuous Glucose Monitoring System

INTERVENTIONS:
Device: Continuous Glucose Monitoring System — The Eversense® 180 CGM System
  Other Names: Eversense CGM system

SUMMARY:
The purpose of this clinical investigation is to evaluate the accuracy of the Eversense® continuous Glucose Monitoring System (Eversense® 180 CGM System) measurements when compared with reference standard measurements up to 180 days of sensor use.

The investigation will also evaluate safety of the Eversense® 180 CGM System usage.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects, age ≥18 years
2. Clinically confirmed diagnosis of diabetes mellitus for ≥1 year
3. Subject has signed an informed consent form and is willing to comply with protocol requirements

Exclusion Criteria:

1. History of unexplained severe hypoglycemia in the previous 6 months. Severe hypoglycemia is defined as hypoglycemia resulting in loss of consciousness or seizure
2. History of diabetic ketoacidosis requiring emergency room visit or hospitalization in the previous 6 months
3. Subjects with gastroparesis
4. Female subjects of childbearing capacity (defined as not surgically sterile or not menopausal for ≥ 1 year) who are lactating or pregnant, intending to become pregnant, or not practicing birth control during the course of the study.
5. A condition preventing or complicating the placement,operation, or removal of the Sensor or wearing of transmitter, including upper extremity deformities or skin condition.
6. Symptomatic coronary artery disease; unstable angina; myocardial infarction, transient ischemic attack or stroke in the past 6 months; uncontrolled hypertension (systolic>160 mm Hg or diastolic >100 mm Hg at time of screening); current congestive heart failure; history of cardiac arrhythmia (benign PACs and PVCs allowed). Subjects with asymptomatic coronary artery disease (e.g. CABG, stent placement or angioplasty) may participate if negative stress test within 1 year prior to screening and written clearance from Cardiologist documented.
7. Hematocrit <30% or >60%
8. History of hepatitis B, hepatitis C, or HIV
9. Current treatment for a seizure disorder unless written clearance by neurologist to participate in study
10. History of adrenal insufficiency
11. Currently receiving (or likely to need during the study period): immunosuppressant therapy; chemotherapy; anticoagulant/antithrombotic therapy (excluding aspirin); glucocorticoids (excluding ophthalmic or nasal). This exclusion does include the use of inhaled glucocorticoids and the use of topical glucocorticoids (over sensor site only); antibiotic for chronic infection (e.g. osteomyelitis, endocarditis)
12. A condition requiring or likely to require magnetic resonance imaging (MRI)
13. Known topical or local anesthetic allergy
14. Known allergy to glucocorticoids
15. Any condition that in the investigator's opinion would make the subject unable to complete the study or would make it not in the subject's best interest to participate in the study. Conditions include but are not limited to psychiatric conditions, known current or recent alcohol abuse or drug abuse by subject history, a condition that may increase the risk of induced hypoglycemia or risk related to repeated blood testing. Investigator will supply rationale for exclusion
16. Participation in another clinical investigation (drug or device) within 2 weeks prior to screening or intent to participate during the study period
17. The presence of any other active implanted device (as defined further in protocol)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2018-12-27 (Actual); Primary Completion 2020-05-08 (Actual); Study Completion 2020-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Satish Garg, MD, Principal Investigator — Barbara Davis Center
Locations (8):
- United States (8):
  - John Muir Physician Network Clinical Research Center, Concord, California
  - AMCR Institute Inc., Escondido, California
  - Diablo Clinical Research, Walnut Creek, California
  - Barbara Davis Center for Diabetes, Aurora, Colorado
  - Atlanta Diabetes Care, Atlanta, Georgia
  - Rocky mountain Diabetes Center C/O Research Department, Idaho Falls, Idaho
  - Clinical Trials of Texas, San Antonio, Texas
  - Rainier Clinical Research Center, Renton, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Continuous Glucose Monitoring Device
Started | 181 (inserted with sensor(s).)
Received SBA Sensor | 43 (43 Subjects received the SBA sensor as a secondary sensor.)
Completed | 171
Not Completed | 10
Not completed — Withdrawal by Subject | 10

BASELINE CHARACTERISTICS:
Population: Subjects enrolled and inserted with the Eversense 180 CGM system.
Groups:
- The Eversense® 180 CGM System All Subject: All subjects inserted with a study sensor(s).
Arm/Group | The Eversense® 180 CGM System All Subject
Number analyzed (Participants) | 181
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96
  Male | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23
  Not Hispanic or Latino | 158
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 163
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 181
Body Mass Index Class [Count of Participants; unit: Participants]
  Normal (<25 kg/m2) | 28
  Overweight (>25 and <30) | 53
  Obese (>30) | 100
Years since diabetes diagnosis [Mean (Standard Deviation); unit: years] | 22.0 (13.3)
Diabetes type [Count of Participants; unit: Participants]
  Type 1 | 126
  Type 2 | 55
Type of insulin therapy [Count of Participants; unit: Participants]
  None (oral diabetes medications only) | 16
  Multiple daily injections | 65
  Continuous insulin infusion pump | 92
  Other (Basal only or 1 injection per day) | 8
History of ketoacidosis and hypoglycemia in past 6 months [Count of Participants; unit: Participants]
  Ketoacidosis | 0
  Hypoglycemia | 0

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness Measure - Mean Absolute Relative Difference (MARD) for Paired CGM and Reference Glucose Measurements
Description: The effectiveness endpoint is the mean absolute relative difference (MARD), calculated for paired CGM Sensor and reference glucose measurements through 180 days post-sensor insertion for reference glucose values from 40-400 mg/dL. MARD is defined as the average of absolute difference of paired Sensor and reference glucose readings divided by the reference glucose reading (reference) for reference glucose values from 40-400 mg/dL, that is: MARD = ((SUM | (Glucose)sensor - (Glucose)reference | / (Glucose)reference ) / n ) x 100%, where n is the total number of Sensor and reference glucose pairs after 180 days of sensor use (MARD is expressed as a percent). Lower MARDs indicate higher (better) accuracy.
Time Frame: 180 days
Measure: Mean (95% Confidence Interval); unit: percent
Units Other Than Participants: Matched CGM and YSI pairs
Groups:
- The Eversense® 180 CGM System All Subject: All subjects inserted with a study sensor
- The Eversense® 180 CGM System SBA Subgroup: Subjects inserted with Eversense® 180 CGM system with slightly modified indicator hydrogel containing sacrificial boronic acid (referred to as SBA Sensor).
Arm/Group | The Eversense® 180 CGM System All Subject | The Eversense® 180 CGM System SBA Subgroup
Number analyzed (Participants) | 181 | 43
Number analyzed (Matched CGM and YSI pairs) | 49613 | 12034
percent | 9.1 [8.7 to 9.5] | 8.5 [8.0 to 9.0]

2. Primary Outcome: Safety Endpoint - Incidence of Device-related or Sensor Insertion/Removal Procedure-related Serious Adverse Events
Description: Incidence of device-related or sensor insertion/removal procedure-related serious adverse events occurring up to 180 days after the insertion procedure.
Time Frame: 180 days
Measure: Number (95% Confidence Interval); unit: serious adverse events
Arm/Group | The Eversense® 180 CGM System All Subject | The Eversense® 180 CGM System SBA Subgroup
Number analyzed (Participants) | 181 | 43
serious adverse events | 0 [0.0 to 2.0] | 0 [0.0 to 8.2]

ADVERSE EVENTS:
Time Frame: Through 180 days post Sensor insertion and sensor removal 10-day follow-up (up to 190 days)
Groups:
- The Eversense® 180 CGM System All Subject Evaluation: All subjects inserted with a study sensor.
Arm/Group | The Eversense® 180 CGM System All Subject Evaluation | The Eversense® 180 CGM System SBA Subgroup
All-Cause Mortality (participants affected / at risk) | 0/181 | 0/43
Serious Adverse Events (participants affected / at risk) | 7/181 | 3/43
Other Adverse Events (participants affected / at risk) | 118/181 | 30/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | The Eversense® 180 CGM System All Subject Evaluation (N=181) | The Eversense® 180 CGM System SBA Subgroup (N=43)
Invasive lobular carcinoma (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Post-surgical staphylococcus infection in left breast (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Humerus Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
hypoglycemic event (Endocrine disorders) | 1 (1) | 0 (0) — This SAE was not related to the device or procedures.
Chronic behavioral issues (Nervous system disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis event requiring hospitalization (Endocrine disorders) | 1 (2) | 1 (2)
hiatal hernia (General disorders) | 1 (1) | 1 (1)
hyperglycemia (Endocrine disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | The Eversense® 180 CGM System All Subject Evaluation (N=181) | The Eversense® 180 CGM System SBA Subgroup (N=43)
Skin irritation, adhesive patch location (including erythema, pruritus, rash, contact dermatitis) (Skin and subcutaneous tissue disorders) | 9 (13) | 2 (4)
Skin irritation, not device related (including abrasion, laceration, redness, tear, rash, contact de (Skin and subcutaneous tissue disorders) | 7 (8) | 1 (1)
Hypopigmentation (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0)
Infection (not related) (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Skin atrophy (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Skin cancer (left forearm, scalp, ear, nose) (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (2)
Infection (insertion/removal site, under adhesive patch) (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Contact dermatitis/Rash (drape adhesive, heat related) (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Burn (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Erythema, insertion site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Seroma, removal site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 28 (31) | 7 (8)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 3 (3)
Influenzas (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (5)
Chest congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chest pain with tachycardia, dizziness (Cardiac disorders) | 1 (1) | 0 (0)
Lower extremity edema, bilateral (Vascular disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Nausea/Vomiting (Gastrointestinal disorders) | 7 (7) | 3 (3)
Abdominal pain/discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (1 w/ dizziness) (Nervous system disorders) | 20 (31) | 4 (5)
Pain (Nervous system disorders) | 9 (10) | 3 (3)
Migraine with nausea (Nervous system disorders) | 1 (1) | 0 (0)
Arm Numbness (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Pain (back, forehead, hand, neck, etc. ) (Musculoskeletal and connective tissue disorders) | 7 (8) | 0 (0)
Muscle/Connective tissue injury (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2)
Bone Fracture (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Sprain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Arthritis/Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (12)
Carpal tunnel (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Trigger finger (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Puncture wound, right foot (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
UTI (Renal and urinary disorders) | 5 (5) | 2 (3)
HSV flare (General disorders) | 1 (1) | 1 (1)
Vaginal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Hyperglycemia/DKA (Endocrine disorders) | 1 (1) | 0 (0)
Hypoglycemic episode (Endocrine disorders) | 2 (3) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Bruising (Blood and lymphatic system disorders) | 13 (22) | 6 (9)
Bleeding (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Iron Deficiency (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Ecchymosis, IV site (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Antibiotic allergy (General disorders) | 1 (1) | 0 (0)
Food/Drink allergy (General disorders) | 1 (1) | 0 (0)
Seasonal allergy (General disorders) | 1 (1) | 0 (0)
Dental work/issues (General disorders) | 8 (8) | 1 (1)
Cataract (Eye disorders) | 4 (6) | 1 (2)
Otitis media (Ear and labyrinth disorders) | 4 (4) | 0 (0)
Sinus infection (Infections and infestations) | 4 (4) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (2) | 0 (0)
Retinopathy (Eye disorders) | 2 (2) | 1 (1)
Cold sores (Infections and infestations) | 1 (1) | 0 (0)
Corneal ulcer (Eye disorders) | 1 (1) | 0 (0)
Lipoplasty, lower extremities (General disorders) | 1 (1) | 1 (1)
Bariatric surgery (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Thumb tip cut off, right (General disorders) | 1 (1) | 0 (0)
Steristrips did not hold, replaced (General disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-04-14): https://cdn.clinicaltrials.gov/large-docs/76/NCT03808376/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-11): https://cdn.clinicaltrials.gov/large-docs/76/NCT03808376/SAP_001.pdf